CLINICAL TRIAL: NCT06253572
Title: Instructional Design and Implementation for Educational Skills Program Based on Constructivist Learning Approach: An Example of Nurse Instructors
Brief Title: Instructional Design and Implementation for Educational Skills Program Based on Constructivist Learning Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ozgul Eycan, Nurse; Lecturer (Istanbul Arel University Nursing Department); PHD Student (IUC- Nursing Education, Doctorate Program), Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IstanbulUC-Nursing-OE-01
Record Dates: First submitted 2024-01-16; First posted 2024-02-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Teacher Training
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Design of the research: This study is a mixed method design. The first part of the study was planned in a quantitative design with a one-group pretest-posttest quasi-experimental type. The second part of the study was planned in qualitative design and phenomenological type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Education
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Educational Skills Program Based on Constructivist Learning Approach
  Instructors need to receive training to improve their teaching skills during their graduate education and after their appointment as instructors. In this study, it is aimed to design and implement an Educational Skills Program based on the Constructivist Learning Approach. The design of the training program was based on the Dick, Carey and Carey (DCC) Instructional Design Model, which is widely known among instructional design models and influenced by constructivism theory. It is aimed that the training skills training program will be carried out by taking adult education into consideration and will be learner-centered. In this study, the training plan is based on the Constructivist Learning Approach 5E model, which is proven to be effective in the literature and widely used. The training program will be conducted through distance education to reach instructors living in different cities and to create common time.

SUMMARY:
A lecturer is a person who, after completing his/her undergraduate education, specializes in the same or a different discipline through postgraduate education and works at a university. The main responsibilities of lecturers are teaching, research, leadership and community service.

The training skills program includes adult education and characteristics of adult learners, basic concepts of education, teaching methods and techniques, instructional technologies, communication skills, curriculum development, implementation and evaluation and aims to improve participants' training skills.

Teaching is among the main responsibilities of lecturers. Instructors need to receive training to improve their teaching skills during their graduate education and after their appointment as instructors. In this study, it is aimed to design and implement an Educational Skills Program based on the Constructivist Learning Approach. The design of the training program was based on the Dick, Carey and Carey (DCC) Instructional Design Model, which is widely known among instructional design models and influenced by constructivism theory. It is aimed that the training skills training program will be carried out by taking adult education into consideration and will be learner-centered. In this study, the training plan is based on the Constructivist Learning Approach 5E model, which is proven to be effective in the literature and widely used. The training program will be conducted through distance education in order to reach instructors living in different cities and to create common time.

DETAILED DESCRIPTION:
A lecturer is a person who, after completing his/her undergraduate education, specializes in the same or a different discipline through postgraduate education and works at a university. The main responsibilities of lecturers are teaching, research, leadership and community service.

The training skills program includes adult education and characteristics of adult learners, basic concepts of education, teaching methods and techniques, instructional technologies, communication skills, curriculum development, implementation and evaluation and aims to improve participants' training skills.

It is recommended to make use of instructional design models in the process of curriculum development. Curriculum design involves determining the ways of teaching in order to create the desired changes in the learner's knowledge and skills. The curriculum to be created in this study was based on the Dick, Carey and Carey (DCC) Instructional Design Model, which is widely known among instructional design models and influenced by constructivism theory. In 2005, Sweetin classified the stages of the model as design, analysis, development and evaluation.

Constructivism is a theory about knowledge and learning. The theory is based on building knowledge from the ground up. The lesson plans in this study will be based on the 5E model developed by Roger Bybee in the 1960s, which is the most preferred constructivist model. The 5E model consists of the following stages: engage-enter, exploration, explanation, elaboration and evaluation.

A review of nursing doctoral curricula in the United States and Canada, which shows that there is insufficient or no course on imparting educational skills, draws attention to this issue. In a study conducted with lecturers working in the department of nursing, it was determined that half of the participants received training on educational skills and almost all of them thought that formation education should be compulsory. In Eycan and Ulupınar's study (2021), it was determined that half of the instructors working in the nursing department received distance education instructor training, and more than half of them needed training on this topic. In the literature, there is a study showing that the online distance education instructor training program positively affected participants' self-efficacy and perceptions of benefit.

Teaching is among the main responsibilities of lecturers. Instructors need to receive training to improve their teaching skills during their graduate education and after their appointment as instructors. In this study, it is aimed to design and implement an Educational Skills Program based on the Constructivist Learning Approach. The design of the training program was based on the Dick, Carey and Carey (DCC) Instructional Design Model, which is widely known among instructional design models and influenced by constructivism theory. It is aimed that the training skills training program will be carried out by taking adult education into consideration and will be learner-centered. In this study, the training plan is based on the Constructivist Learning Approach 5E model, which is proven to be effective in the literature and widely used. The training program will be conducted through distance education in order to reach instructors living in different cities and to create common time.

Aim of the research:

In this study, it is aimed to develop a distance education program to improve the educational skills of instructors working in departments providing nursing education. Educational skills training will be carried out by distance education in order to reach instructors living in different cities and to create common time. The training program will be created in line with the Dick, Carey and Carey Instructional Design Model. Lesson plans will be based on the Constructivist Learning Approach 5E model. As a result of the study, it is aimed to provide the nursing literature with a distance education program for educational skills based on the 5E model. It is thought that it can be applied by other departments in higher education by making minimal edits in the education program to be developed.

Design of the research:

This study is a mixed method design. The first part of the study was planned in a quantitative design with a one-group pretest-posttest quasi-experimental type. The second part of the study was planned in qualitative design and phenomenological type.

Hypothesis:

H1: The mean score of the Educational Skills Scale of the nurse lecturers participating in the Educational Skills Program Based on Constructivist Learning Approach 3 months after the theoretical training is higher than before the training.

H2: Educational Skills Program Based on Constructivist Learning Approach is an effective training program.

Research questions:

Did the average scores of the teaching staff on the Training Skills Scale increase after the training? What are the factors affecting the training skills of the instructors? Is there a significant difference in the evaluation of the presentations organized in the practice phase of the training by self, peer and educator? What are the opinions of the participants about the training program? What is the contribution of the program to the participants' educational skills?

Participants:

The population of the study will consist of lecturers working in the Nursing Departments of universities in Turkey. Priority will be given to research assistants among the lecturers. In determining the sample size, a calculation was made using the mean and standard deviation values in a study examining the educational skills of nurse lecturers. GPOWER 3.1 package program was used in sample calculation. According to the GPOWER analysis, the minimum sample size to ensure the power of the test (1-β) = 0.80 was determined as 27 by taking the Type 1 margin of error (α) 0.05.

Sampling inclusion criteria:

Graduating from the Department of Nursing. To be enrolled in or graduated from a master's or doctoral program in one of the departments of nursing.

To be working as a lecturer in nursing departments. In the study, priority will be given to those working as research assistants in nursing departments.

Priority will be given to those who have been working as a lecturer in the nursing department for a maximum of 2 years.

Priority will be given to those who have given and continue to give theoretical or laboratory or application courses in the nursing department.

In the qualitative part of the study, it was planned to conduct individual in-depth interviews with a randomly selected group of those who completed the training program and volunteered to participate in the interview.

Sampling exclusion criteria:

Becoming a faculty member, Not having a nursing degree, Graduate education in a field other than one of the nursing departments

Data collection:

The forms to be used in the quantitative part of the study are listed below. Information Form: The form was created by the researcher by reviewing the relevant literature.

Education Skills Scale: The scale developed by Çayır and Ulupınar (2021) consists of a total of 38 items and is a five-point Likert scale (1. Never, 2. Rarely/Sometimes, 3. Sometimes/Sometimes, 4. Often/Frequently, 5. Always). All statements in the scale are positive. Each item in the scale is given a score between 1-5. The minimum score is 38 and the maximum score is 190. It was determined that the higher the score obtained from the Training Skills Scale, the higher the frequency of using training skills. The Cronbach Alpha coefficient of the scale was determined to be 0.93.

Scale On Assessing Constructivist Learning Environment: The scale developed by Arkün and Aşkar in 2010 is a seven-point Likert scale (1 strongly disagree to 7 strongly agree). The scale consists of 28 items and six factors: student-centered, thought-provoking, collaborative, life-related, teaching and evaluation together, and providing different perspectives.

Presentation evaluation form: The "Presentation Evaluation Form" was prepared by the researchers to evaluate the presentations to be made during the practice phase of the training. The form consists of 10 items. The form was prepared as a rubric. Each item will be scored as "Not done" 0, "Inadequate" 1, "Needs improvement" 2 and "Adequate" 3. Participants will be able to get a score between 0 and 30 points from the form. The higher the score obtained from the form, the higher the presentation skill will be accepted.

The form to be used in the qualitative part of the study are listed below. In the qualitative dimension of the study, individual in-depth interviews will be conducted with a randomly selected group of participants and their opinions on the training program and their achievements related to the training program will be obtained. A semi-structured interview form will be used in the interviews and the draft of the form was created by the researcher by examining the relevant literature.

Data Collection Methods:

In the quantitative part of the study, data will be collected online with Google forms and in the qualitative part of the study, data will be collected on platforms such as online zoom.

Ethical considerations:

Ethics committee permission for the study was obtained from Istanbul Arel University Ethics Committee with the board decision dated 28/04/2023 and numbered 2023/09. The permission to use the scales to be used in the study was obtained from the researchers who developed the scale. Data will be collected online. Therefore, permission was not obtained from any institution. Participants will be sent an informed consent form explaining the purpose and process of the study. Participants who give consent will be included in the study.

Data Analysis:

In the quantitative part of the study, the analysis of the data will be evaluated with the Statistical Package for Social Sciences (SPSS) 24.0 Windows program and the statistical significance value will be accepted as p<0.05 in the analysis. Appropriate statistical analyzes will be used to analyze the data.

In the qualitative part of the study, it is planned to use the thematic analysis method to analyze the data.

This study is a doctoral thesis.

ELIGIBILITY:
Inclusion Criteria:

* Graduating from the Department of Nursing.
* To be enrolled in or graduated from a master's or doctoral program in one of the departments of nursing.
* To be working as a lecturer in nursing departments.
* In the study, priority will be given to those working as research assistants in nursing departments.
* Priority will be given to those who have been working as a lecturer in the nursing department for a maximum of 2 years.
* Priority will be given to those who have given and continue to give theoretical or laboratory or application courses in the nursing department.
* In the qualitative part of the study, it was planned to conduct individual in-depth interviews with a randomly selected group of those who completed the training program and volunteered to participate in the interview.

Exclusion Criteria:

* Becoming a faculty member,
* Not having a nursing degree,
* Graduate education in a field other than one of the nursing departments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Education Skills Scale | up to 12 months
  Education Skills Scale: The scale developed by Çayır and Ulupınar consists of a total of 38 items and is a five-point Likert scale (1. Never, 2. Rarely/Sometimes, 3. sometimes/ Sometimes, 4. Often/Frequently, 5. Always). All statements in the scale are positive. Each item in the scale is given a score between 1-5. The minimum score is 38 and the maximum score is 190. It was determined that the higher the score obtained from the Training Skills Scale, the higher the frequency of using training skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Unıvercity- Cerrahpasa, Avcılar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bullin C. To what extent has doctoral (PhD) education supported academic nurse educators in their teaching roles: an integrative review. BMC Nurs. 2018 Feb 22;17:6. doi: 10.1186/s12912-018-0273-3. eCollection 2018. PMID 29483844
- [Result] Eycan O, Ulupinar S. Nurse instructors' perception towards distance education during the pandemic. Nurse Educ Today. 2021 Dec;107:105102. doi: 10.1016/j.nedt.2021.105102. Epub 2021 Aug 18. PMID 34482209
- [Result] Cayir A, Ulupinar S. The relationship among educational skills, general self-efficacy perceptions and performance in nursing instructors. Nurse Educ Today. 2021 Dec;107:105129. doi: 10.1016/j.nedt.2021.105129. Epub 2021 Sep 2. PMID 34534784
- Available data/document: Individual Participant Data Set — http://dergipark.org.tr/en/pub/auad/issue/60075/826745
- Available data/document: Review — http://dergipark.org.tr/en/download/article-file/411491
- Available data/document: Review — http://journalofomepturkey.org/index.php/eccd/article/view/78
- Available data/document: master's thesis — http://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp — Tahta, N. (2022). Creation of a program for training of military trainers. (Unpublished master's thesis). İstanbul: National Defence University.
- Available data/document: Review — http://dergipark.org.tr/en/download/article-file/199140
- Available data/document: Individual Participant Data Set — http://dergipark.org.tr/en/pub/rep/issue/63330/827844